CLINICAL TRIAL: NCT01354288
Title: Therapeutic Education in Very Young Children With Diabetes Mellitus. Evaluation of the Impact of a Specific Tool for Parents on Glycemic Control and Prevention of Acute Events (Hypoglycemia and Ketosis)
Brief Title: Therapeutic Education in Very Young Children With Diabetes Mellitus
Acronym: DIAB-EDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P081254
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus
Keywords: Diabetes; Children; Disease management; Ketosis; Hypoglycemia; Parents; Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Ketosis; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education (Experimental)
  Interventions: Other: Educational tool
- Classical management (No Intervention)

INTERVENTIONS:
Other: Educational tool — Specific educational tool in order to assess its impact on glycemic control, quality of life, knowledge about the disease and its daily management
  Other Names: Experimental
  Arms: Therapeutic education

SUMMARY:
DIAB-EDUC tests in a group of young diabetic patients (less than 6 years old) a specific educational tool in order to assess its impact on glycemic control, quality of life, knowledge about the disease and its daily management, over a period of 2 years. The investigators plan to include 300 type 1 diabetic children in 10 french hospitals.

DETAILED DESCRIPTION:
General frame : 1 inclusion / randomization visit and delivery of the educational tool for patients of the "Therapeutic Education" arm, then follow-up visits every 6 months during 24 months.

V0 - Inclusion / randomization visit - Verification of eligibility - Clinical examination and data report - Blood samples for lab tests (HbA1c assay)- Collection of signed consent form- DIAB-EDUC questionnaire (diabetes knowledge, treatment, quality of life, hypoglycaemia and emergency situations, parental stress)- Randomization - Education tool explanation and delivery by the physicians to parents randomized in " Experimental " arm

M6 - Visit at 6 months- Clinical examination and data report- Blood samples for lab tests (HbA1c assay)

M12 - Visit at 12 months- Clinical examination and data report- Blood samples for lab tests (HbA1c assay)- DIAB-EDUC questionnaire

M18 - Visit at 18 months- Clinical examination and data report- Blood samples for lab tests (HbA1c assay)

M24 - Visit at 24 months- Clinical examination and data report- Blood samples for lab tests (HbA1c assay)- DIAB-EDUC questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Children with type 1 diabetes aged 1 to 6 years
* Disease evolution more than 1 year
* HbA1c > 8% or at least one acute accident (hypoglycemia or ketosis) during the last year
* Specific information given to parents from the physicians and consent form signed by the parents
* Physical examination of the children at enrolment- patient affiliated with or receiving health insurance

Exclusion Criteria:

* Non-insulin dependent diabetes
* Monogenic diabetes (MODY)
* Severe co-morbidities- cognitive disabilities or psychosocial disadvantage compromising the therapeutic education
* Children whose parents have a disorder of comprehension or expression of the French Language
* Patients included in another interventional trial

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
HbA1c 12 months after therapeutic education | 12 months

SECONDARY OUTCOMES:
HbA1C 24 months after therapeutic education | 24 months
Acute events number (hypoglycemia and ketosis) over a 12 and 24 months period | 12 and 24 months
Evolution of the parental knowledge about the disease 12 and 24 months after therapeutic education (evaluated by questionnaire) | 12 and 24 months
Evolution of the parental stress 12 and 24 months after therapeutic education (evaluated by questionnaire) | 12 and 24 months
Evolution of the parental and child quality of life 12 and 24 months after therapeutic education (evaluated by questionnaire) | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUGNERES, MD, PhD, Principal Investigator — Bicêtre Hospital
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France